CLINICAL TRIAL: NCT00492713
Title: Comparison of the Bioavailability of Polyphenols From Milk and Dark Chocolate
Brief Title: Polyphenol Bioavailability From Chocolate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 06.31.MET
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: Bioavailability; Dark Chocolate; Milk Chocolate; Polyphenols

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Dark chocolate
  Interventions: Other: dark chocolate
- 2 (Active Comparator): Milk chocolate 1
  Interventions: Other: Milk chocolate 1
- 3 (Active Comparator): Milk chocolate 2
  Interventions: Other: Milk chocolate 2

INTERVENTIONS:
Other: dark chocolate — dark chocolate
  Arms: 1
Other: Milk chocolate 1 — Milk chocolate 1
  Arms: 2
Other: Milk chocolate 2 — Milk chocolate 2
  Arms: 3

SUMMARY:
Dark chocolate is one of the richest sources of polyphenols though it has been hypothesised that the bioavailability of epicatechin from milk chocolate was reduced compared to dark. The primary outcome measure is to compare plasma polyphenol levels after consumption of 3 chocolates (2 milk, 1 dark) while the secondary outcome measures are to characterise the time course of polyphenols in the blood and to investigate individual variation in Tmax and Cmax for use in future studies.

DETAILED DESCRIPTION:
Dark chocolate is one of the richest sources of polyphenols, for example, a standard 40g portion of dark chocolate contains 400-800 mg of polyphenols, compared to red wine (170 mg /100ml) or an apple (200 mg/piece). Cocoa polyphenols, most notably the catechins, can exist in both lipid and water-based environments (amphipathic), meaning they can spare both lipophillic and hydrophilic vitamins. There have been a number of human trials conducted using chocolate or cocoa and measuring various endpoints. Most have been conducted with dark chocolate. An article in Nature found that the bioavailability of epicatechin from milk chocolate was substantially reduced compared to dark, and even dark taken with a glass of milk (Serafini et al 2003). The hypothesis was that the milk proteins bind to polyphenols, making them unavailable. Subsequent studies have not been able to reproduce this, but none have been conducted using solid chocolate as the first study, all have been done using a drink matrix, which may completely alter the binding interactions of the polyphenols and protein. Previous bioavailability trials with dark chocolate have shown a 12 fold increase in plasma epicatechin 2 hours after consumption of 80g of chocolate containing 557 mg total polyphenols (137 mg epicatechin) (Rein et al 2000) with a concurrent increase in plasma total antioxidant capacity and a decrease in TBARS. Another study showed an increase in epicatechin 2 hours after administering 25g of chocolate chips containing 220 mg flavanols and procyanidins, with a concurrent increase in prostacyclin/leukotriene ratio and reduction in platelet-related hemostasis (Holt et al 2002).

This study is designed as a blinded, three arm crossover trial. The primary outcome measure is to compare plasma polyphenol levels after consumption of 3 chocolates (2 milk, 1 dark) while the secondary outcome measures are to characterise the time course of polyphenols in the blood and to investigate individual variation in Tmax and Cmax for use in future studies. All volunteers will try all chocolate types with a similar taste & appearance (though milk and dark are likely to still be distinguishable for the volunteer, not the investigator). Subjects will undergo medical screening, anthropometry, physical activity and dietary assessments before randomisation for the order of consumption. Bloods are to be taken as a time course for the next 24 hours, as is urine.

ELIGIBILITY:
Inclusion Criteria:

* 19 - 45 years, male and female
* Healthy as determined by the medical questionnaire
* Normal weight: BMI 19 - 25
* Having given informed consent

Exclusion Criteria:

* Intestinal or metabolic diseases/disorders such as diabetic, renal, hepatic, hypertension, pancreatic or ulcer, including lacto-intolerance.
* Have had a major gastrointestinal surgery.
* Have a regular consumption of medication.
* Have an exceptionally high intake of chocolate or similarly high polyphenol foods.
* Have a high and regular intake of vitamin supplements
* Have an alcohol intake: > 2 units a day
* Patient who cannot be expected to comply with treatment.
* Smoker
* Having a nut allergy
* Unwilling to consume chocolate
* Currently participating or having participated in another clinical trial during the last 3 weeks.
* Having given blood in the past three weeks
* More than 3 x 45 min of exercise per week

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-06; Primary Completion 2008-09 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
AUC plasma polyphenols | 24 hours

SECONDARY OUTCOMES:
Tmax and Cmax of plasma polyphenols | 24 hours
Plasma and urinary metabolite identification and quantification | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Karen A Cooper, PhD, Principal Investigator — Société des Produits Nestlé (SPN); Gary Williamson, PhD, Study Director — Société des Produits Nestlé (SPN)
Locations (1):
- Nestle Research Center, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Serafini M, Bugianesi R, Maiani G, Valtuena S, De Santis S, Crozier A. Plasma antioxidants from chocolate. Nature. 2003 Aug 28;424(6952):1013. doi: 10.1038/4241013a. No abstract available. PMID 12944955